CLINICAL TRIAL: NCT00000974
Title: A Phase I Study of the Safety, Tolerance, and Study of the Pharmacokinetics of Aerosolized Pentamidine and Parenteral Pentamidine in Children With HIV Infection and Suspected Pneumocystis Carinii Pneumonia
Brief Title: A Study of Two Forms of Pentamidine in HIV-Infected Children Who May Have Pneumocystis Carinii Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 115; 11090 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Injections, Intravenous; Drug Evaluation; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate the delivery of a single dose of aerosolized pentamidine to children; to evaluate the tolerance of pentamidine administration by mask; to compare intravenous pentamidine first dose pharmacokinetics (blood levels) in children with information previously collected on adults; and to compare plasma pentamidine levels in children after an aerosolized treatment with levels previously collected on adults.

Pneumocystis carinii pneumonia (PCP) is the most common serious infection in children with AIDS and is associated with a high death rate. Current approved treatment includes intravenous trimethoprim - sulfamethoxazole (TMP / SMX) and intravenous pentamidine, which are both effective in treatment of the first episode of PCP pneumonia. However, both therapies have a 50 percent or greater incidence of adverse reactions. Because of serious toxicities, drug treatment has had to be discontinued. Animal studies show that aerosolized pentamidine (pentamidine given through inhalation) is as effective as intravenous pentamidine. It is hoped that the aerosolized route will be less toxic than intravenous pentamidine. The study is the first step in evaluating the delivery of aerosolized pentamidine to children.

DETAILED DESCRIPTION:
Pneumocystis carinii pneumonia (PCP) is the most common serious infection in children with AIDS and is associated with a high death rate. Current approved treatment includes intravenous trimethoprim - sulfamethoxazole (TMP / SMX) and intravenous pentamidine, which are both effective in treatment of the first episode of PCP pneumonia. However, both therapies have a 50 percent or greater incidence of adverse reactions. Because of serious toxicities, drug treatment has had to be discontinued. Animal studies show that aerosolized pentamidine (pentamidine given through inhalation) is as effective as intravenous pentamidine. It is hoped that the aerosolized route will be less toxic than intravenous pentamidine. The study is the first step in evaluating the delivery of aerosolized pentamidine to children.

Sixteen patients are assigned into one of the following groups. Group 1 (four patients) receives intravenous pentamidine as a one-time dose, infused over 2 hours. Group 2a (six patients) receives aerosolized pentamidine via face mask. Group 2b (six patients) receives aerosolized pentamidine 2 times. Group 2b will be studied only if initial dose is well tolerated. Small amounts (1 - 2 cubic centimeters) of blood is taken from all groups at 40 minutes, and 2, 3, 7, 14, and 24 hours from the beginning of pentamidine treatment and at the same time as the lung biopsy or bronchial alveolar lavage. Patients are given routine TMP / SMX (or whatever medications are considered appropriate by the patient's primary physician for medical management) dosing 1 - 2 hours after pentamidine is given. Bronchial alveolar lavage fluid or lung tissue from biopsy will be obtained between 2 - 48 hours after initiation of pentamidine treatment (optionally 10 - 24 hours post dose).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Routine trimethoprim / sulfamethoxazole (TMP / SMX) (or whatever medications are considered appropriate by the patient's primary physician for medical management) 1 - 2 hours after pentamidine is given.

Patients must have:

* HIV infection with suspected Pneumocystis carinii pneumonia (PCP).
* Parent(s) or legal guardian must sign an informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Known history of reactive airway disease or another chronic lung disease.
* Known previous adverse reaction to pentamidine.
* Thrombocytopenia.

Patients with the following are excluded:

* History of reactive airway disease or another chronic lung disease.
* Known previous adverse reaction to pentamidine.

Unable to cooperate with administration of aerosol via face mask.

Ages: 2 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: YJ Bryson, Study Chair; ER Stiehm, Study Chair; B Montgomery, Study Chair
Locations (4):
- United States (4):
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Texas Children's Hosp. CRS, Houston, Texas

REFERENCES:
- [Background] Conte JE Jr; Wara D. Pharmacokinetics of aerosolized pentamidine in children. Int Conf AIDS. 1993 Jun 6-11;9(1):381 (abstract no PO-B10-1477)
- [Background] Kreuz W, Gunguor T, Funk M, Ehrenforth S, Linde R, Lotz C, Kornhuber B. First experience with Pneumocystis carinii pneumonia-prophylaxis by inhaled pentamidine in HIV-infected children. Int Conf AIDS. 1991 Jun 16-21;7(2):242 (abstract no WB2243)